CLINICAL TRIAL: NCT04264351
Title: Frailty, Anesthesia and Complications in an Urological Setting.
Brief Title: Frailty, Anesthesia and Complications.
Acronym: FRAC
Status: Completed | Type: Observational
Sponsor: Fundacio Puigvert (Other)
Collaborators: Parc Sanitari Pere Virgili (Other)
Responsible Party: Principal Investigator, Merce Prieto Butillé, MD, Anesthesiology consultant, Fundacio Puigvert
Other Study IDs: FRAC1
Record Dates: First submitted 2019-01-03; First posted 2020-02-11 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Frail Elderly Syndrome; Anesthesia Complication; Complication of Surgical Procedure; Postoperative Delirium; Physical Disability
Keywords: Frailty; Anesthesia; complications
MeSH Terms: conditions — Emergence Delirium; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objectives: To assess the prevalence of frailty in patients older than 70 y/o in nephrourologic surgery. To study if preoperative frailty is an independent predictor of immediate postoperative complications, after 30 days, 6 months and 1 year of follow-up. To detect if there are other independent risk factors for complications.

DETAILED DESCRIPTION:
Objectives: To assess the prevalence of frailty in patients older than 70 y/o in nephrourologic surgery. To study if preoperative frailty is an independent predictor of immediate postoperative complications, after 30 days, 6 months and 1 year of follow-up. To detect if there are other independent risk factors for complications.

Methods: prospective cohort study performed at Fundació Puigvert. Enrollment of 850 patients ≥70 y/o who undergo scheduled nephrourologic surgery. In the preoperative visit frailty is going to be evaluated using the Short Physical Performance Battery (SPPB), the Canadian Frailty Scale, the Mini-Cog test (Memory an executive functions), the Pfeiffer Test (Cognitive global screening), an involuntary loss of more than 4.5kg or 5% of weight in the previous year and physical activity using the Metabolic Equivalents of Task (MET). We will analyse the relation among frailty, medical, surgical postoperative complications and mortality at 30 days, 6 months and one year after the surgery.

The results will be adjusted by the possible confounding and interaction variables using a multivariate logistic regression model. The confounding /interaction variables will include demographic data, clinical and lab data and events arisen during the follow-up period.

ELIGIBILITY:
Inclusion criteria

* Patients who participate voluntarily
* Signed Informed consent
* 70+ years old
* Scheduled urological surgery with general or regional anesthesia and length of stay in hospital over 24 hours.
* Patients with preserved domiciliary deambulation without aid of another person. (walking sticks, or walkers are accepted)

Exclusion Criteria:

* No signing of the informed consent
* Surgery performed with local anesthetics
* Day surgery, extracorporeal wave lithotripsy or endourological catheterism
* Advanced diagnosed dementia
* Patients with chronic advanced disease or terminal oncological disease

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing urological scheduled surgery in our centre, that fill in the inclusion criteria with no exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Frailty as a risk factor of postoperative events. | 2017-2021
  Assessment the prevalence of frailty in the surgical settings defined as a clinically recognizable state of increased vulnerability resulting from aging-associated decline in reserve and function across multiple physiologic systems. Frailty is defined as meeting three out of five phenotypic criteria indicating compromised energetics: low grip strength, low energy, slowed waking speed, low physical activity, and/or unintentional weight loss
Frailty will be evaluated during the preoperative visit of patients 70+ scheduled to uronephrologic surgery | 2017-2021
  Frailty is going to be evaluated in the anesthetic preoperative visit using the Short Physical Performance Battery (SPPB), Canadian Frailty Scale, Mini-Cog test (Memory an executive functions), Pfeiffer Test (Cognitive global screening), Involuntary loose of more than 4,5kg or 5% of weight in the previous year, physical activity using the Metabolic Equivalents of Task (MET).

SECONDARY OUTCOMES:
Postoperative events and frailty | 2017-2021
  Assessment of the association among frailty, medical and surgical postoperative complications at 30 days, 6 months and one year after the surgery.
Mortality associated to frailty and its complications | 2017-2021
  Assessment of the association between frailty and mortality at 30 days, 6 months and one year after the surgery.
Preoperative visit as a chance to assess frailty | 2017-2021
  Analyze which frailty evaluation tool works better in the preoperative visit setting.

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Sabate, MD PhD, Study Director — Chair Anesthesiologist at Fundació Puigvert
Locations (1):
- Fundació Puigvert, Barcelona, Spain